CLINICAL TRIAL: NCT05090150
Title: A Sequential Multiple Assignment Randomized Trial of Scalable Interventions for ART Delivery in South Africa: the SMART ART Study
Brief Title: The SMART ART Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ruanne Barnabas, MBChB, MSc, DPhil., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P001129; R01MH124465 (NIH)
Record Dates: First submitted 2021-09-16; First posted 2021-10-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV; ART

STUDY DESIGN:
Intervention Model Description: Participants are first randomly assigned to two interventions:either best clinic practices or best clinic practices with a conditional lottery incentive. This stage lasts 6 months. Participants who do not meet the criteria for non-response will continue in the assigned intervention arm. Non-responders will be rerandomized to continue in the clinic intervention arm (standard of care), community ART (smart lockers), or home delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Best clinic practices (No Intervention): Participants start with best clinic practices and continue for 18 months (including participants who are non-responders at month 6 and are randomized to stay in their original arm)
- Best clinic practices plus lottery incentives (Experimental): Participants start with best clinic practices plus lottery incentives and continue for 18 months (including participants who are non-responders at month 6 and are randomized to stay in the original arm)
  Interventions: Other: Best clinic practices + conditional lottery incentives
- Randomized from best clinic practices to smart lockers (Experimental): Second randomization into community ART through the use of smart lockers
  Interventions: Other: Smart Lockers (Pele boxes); Other: Best clinic practices
- Randomized from best clinic practices to home delivery (Experimental): Second randomization into home ART delivery
  Interventions: Other: Home delivery of ART; Other: Best clinic practices
- Randomized from best clinic practices plus lottery incentives to smart lockers (Experimental): Second randomization into community ART through the use of smart lockers
  Interventions: Other: Smart Lockers (Pele boxes); Other: Best clinic practices + conditional lottery incentives
- Randomized from best clinic practices plus lottery incentives to home delivery (Experimental): Second randomization into home ART delivery
  Interventions: Other: Home delivery of ART; Other: Best clinic practices + conditional lottery incentives

INTERVENTIONS:
Other: Home delivery of ART — Home ART refill and monitoring, adherence support
  Arms: Randomized from best clinic practices plus lottery incentives to home delivery; Randomized from best clinic practices to home delivery
Other: Smart Lockers (Pele boxes) — Decentralized ART refills and monitoring, adherence support
  Arms: Randomized from best clinic practices plus lottery incentives to smart lockers; Randomized from best clinic practices to smart lockers
Other: Best clinic practices + conditional lottery incentives — Conditional lottery incentives Welcome back service (friendly providers, SMS, adherence support) Fast-track ART
  Arms: Best clinic practices plus lottery incentives; Randomized from best clinic practices plus lottery incentives to home delivery; Randomized from best clinic practices plus lottery incentives to smart lockers
Other: Best clinic practices — Continue with best clinic practices
  Arms: Randomized from best clinic practices to home delivery; Randomized from best clinic practices to smart lockers

SUMMARY:
The investigators propose A Sequential Multiple Assignment Randomized Trial of scalable interventions for ART delivery in South Africa- the SMART ART study-a randomized study to test adaptive ART delivery for persons with detectable viral load and/or not engaged in care.The types of differentiated service delivery (DSD) that will be examined in this study are incentives, community-based ART, and home delivery. The study plans to enroll up to 900 participants-people living with HIV and who are eligible for ART and living in KwaZulu-Natal, South Africa. The study aims to maximize the proportion of ART eligible persons living with HIV who achieve viral suppression at 18 months. The study will also evaluate the preferences of clients and providers for differentiated service delivery, and evaluate the cost effectiveness of adaptive HIV treatment for those who are not engaged in care.

DETAILED DESCRIPTION:
Of the 8 million people in South Africa living with HIV, only 56% are on antiretroviral therapy (ART), and 45% are virally suppressed, substantially below the UNAIDS goal of 73%. Detectable viral load results in HIV-associated morbidity and mortality, and HIV transmission. Patient barriers to care, such as missed wages, transport costs, and long wait times for clinic visits and ART refills, are associated with detectable viral load. HIV differentiated service delivery (DSD) has simplified ART delivery: incentives, multi-month scripts, fast-track ART, and community or home ART delivery motivate clients, reduce the frequency of clinic visits, and decongest clinics. DSD is standard for clients who achieve viral suppression and engage in care; however, DSD needs adaptation to serve clients who are not succeeding. Indeed, persons who are not engaged in care arguably need simplified, client-centered approaches even more than those who can successfully engage.

A suite of adaptive DSD strategies, including incentives strategies, community-based ART, and home delivery, have been tested among stable clients with viral suppression. Lottery incentives effectively change short-term behavior, increasing ART initiation.Community-based and home ART delivery increase ART coverage and simplify ART access overcoming clinic barriers11. For stable clients, these DSD activities are as effective as clinic-based care in terms of achieving and maintaining viral suppression, although among stable clients they have not shown superiority in viral suppression or cost savings. In contrast, DSD has the potential to improve rates of viral suppression and retention in care and save costs among persons not engaged in care. There is great potential that DSD systems can be client-responsive and system-efficient for subgroups requiring additional services, matching services with client needs. A sequential, comprehensive package of DSD approaches, with each step increasing the intensity of service provision - adaptive DSD - has not been tested to determine the proportion and characteristics of persons who would achieve viral suppression and retention in care and to estimate the cost-effectiveness and budget impact.

To increase population level viral suppression, persons with detectable viral load need responsive DSD interventions. A Sequential Multiple Assignment Randomized Trial (SMART) design facilitates evaluation of a stepped, adaptive approach to achieving viral suppression with 'right-sized' interventions. The investigators are an experienced team and propose to build on the strong partnerships to sequentially test adaptive DSD strategies for persons with detectable viral load and/or not engaged in care: incentives, community-based ART, and home delivery. As the Center for Community Based Research, the investigators maintain strong connections with stakeholders including department of health, traditional leaders and ward counsellors throughout the Greater Edendale Area (GEA) and the Vulindlela sub-district of the uMgungundlovu District Municipality. Due to the size of the recruitment target, this work will centre around the Caluza clinic but will extend into other parts of GEA and sub-district of Vulindlela over the course of recruitment. The aim is to identify the most effective and efficient HIV care delivery strategies.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Able and willing to provide informed consent for study procedures
* Must self report that they will reside in the study community for the duration of follow-up
* Living with HIV and eligible for ART by national guidelines, have a detectable viral load greater than the lower limit of detection and/or not engaged in care, and are stable clinically (CD4>100 cells, no moderate/severe screening laboratory abnormalities for kidney function i.e. eGFR >50 mL/min/1.73m2, not receiving treatment for active tuberculosis or other opportunistic infections).

Exclusion Criteria:

* There are no separate exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 874 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Viral suppression at 18 months | 18 months
  The primary outcome is viral suppression at 18 months among the combined group of persons living with HIV who have detectable viral load and persons not engaged in care at enrollment.

SECONDARY OUTCOMES:
Retention in Care | 12 months
  The proportion of clinical visits and medication refills missed over the last 12 months of the intervention
Time to ART initiation | 6 months
  Time to antiretroviral therapy initiation
Engagement in care | 18 months
  Proportion of people who are virally suppressed in each intervention arm
Comparison to viral suppression and retention outcomes from similar local clinics | 18 months
  Proportion of individuals who are virally suppressed who are engaged in care in intervention arms compared to local clinics

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne V Barnabas, DPhil, Principal Investigator — University of Washington
Locations (1):
- Human Sciences Research Council Sweetwaters, Sweetwaters, KwaZulu-Natal, South Africa

REFERENCES:
- [Result] van Heerden A, Szpiro A, Ntinga X, Celum C, van Rooyen H, Essack Z, Barnabas R. A Sequential Multiple Assignment Randomized Trial of scalable interventions for ART delivery in South Africa: the SMART ART study. Trials. 2023 Jan 17;24(1):32. doi: 10.1186/s13063-022-07025-x. PMID 36647092